CLINICAL TRIAL: NCT02647671
Title: The Effects of Calcium in Conjunction With Multi-mineral Supplementation (Aquamin) on Gut Microbes and Microbially-derived Metabolites in Subjects at Risk for Colon Cancer in a Randomized Controlled Trial
Brief Title: Aquamin and Prevention of Colon Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James Varani (Other)
Responsible Party: Sponsor-Investigator, James Varani, Professor of Pathology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HUM00076276
Record Dates: First submitted 2015-11-30; First posted 2016-01-06 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Colonic Cancer
Keywords: Colon polyp; Colorectal cancer; Chemoprevention; Natural product
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps; Colorectal Neoplasms | interventions — Aquamin; Calcium Carbonate; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aquamin® (Experimental): Experimental: Aquamin® (4 capsules per day) - 4 capsules; 2 to be taken in the morning and 2 in the evening
  Interventions: Drug: Aquamin®
- Calcium Carbonate (Active Comparator): Active Comparator: Calcium Carbonate (4 capsules per day) - 4 capsules; 2 to be taken in the morning and 2 in the evening
  Interventions: Drug: Calcium Carbonate
- Placebo (Placebo Comparator): Placebo (Maltodextrin) - 4 capsules; 2 to be taken in the morning and 2 in the evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aquamin® — 90 days of Aquamin
  Arms: Aquamin®
Drug: Calcium Carbonate — 90 days of Calcium Carbonate
  Arms: Calcium Carbonate
Drug: Placebo — 90 days of placebo
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
In the proposed study, investigators will conduct a 90-day dietary intervention study in human subjects. Thirty individuals at risk for adenomatous colon polyp formation will be randomized to receive a calcium and multi-mineral-rich natural product (Aquamin) or a comparable level of calcium alone. There will also be a placebo group. Prior to ingesting the study agents and following the course of treatment, colonic biopsies will be obtained by sigmoidoscopy and quantitatively examined for markers of growth and differentiation. In this study, metabolomic and microbial profiles will also be generated from fecal and colon mucosal samples taken at baseline and study endpoint.

DETAILED DESCRIPTION:
The purpose of this study is to see what effects a calcium-rich, multi-mineral-rich natural product, Aquamin®, derived from marine algae, has compared to calcium alone or a sugar pill (placebo). Investigators are looking at whether these supplements do anything to the cell lining of the colon. Specifically, to see if Aquamin®, calcium, or placebo (sugar pill) change markers of cell growth and differentiation (or "biomarkers") in the cells of the colon. The natural product, Aquamin®, contains calcium but, in addition, has a significant amount of magnesium and measurable levels of approximately 70 different trace elements (essentially, everything the algae can accumulate from seawater). Aquamin is a product that is marketed for the fortification of food, beverage, and supplement products. In this study, it is being used for research and therefore, its use is investigational. Calcium supplements have been shown to reduce colonic polyps (precursor lesions to colon cancer). This study will NOT look at polyp formation in the colon, but only at biomarkers of colon cell growth and function. If investigators find that the multi-mineral natural product is substantially more effective than calcium alone in changing these biomarkers, it is possible that a larger study could be conducted that is intended to study colon polyp prevention. In order to test these ideas investigators need to compare the supplement Aquamin®, to something already tested (calcium) and a placebo (sugar pill) to see if any changes are related to the supplements or just naturally happen.

There is increasing recognition that dietary or environmental predispositions to colorectal cancer may be mediated at least in part by alterations of gut microbial composition and metabolomic profiles. Human gut microbiota are now recognized to play an important role in host health and changes in the composition of gut microbial communities have been linked with metabolic alterations that affect colorectal cancer risk. Investigators have previously established that dietary supplementation can correlate with metabolic or microbial alterations in their most recent long-term study in mice on high-fat western diet (HFWD) and calcium. Investigators had also demonstrated that Aquamin-supplemented mice had significantly decreased liver and colon tumors. Based on these studies, investigators anticipate that Aquamin will improve the gut microbial composition and alter the metabolomic profile in these subjects.

If participant agree to participate in this research study, he/she will be asked to sign this informed consent document before any tests are performed or data collected. This research study consists of three time periods (phases): a pre-treatment period; a study treatment period; and an end-of-study treatment period. The study requires three visits to the University of Michigan's Clinical Research Unit (MCRU). These are referred to as the Screening Visit, Baseline Visit and Final Visit.

After participants are determined to meet eligibility requirements, they will be randomized as to which product they will receive. Randomization is like a flip of a coin. A participant will have an equal chance (33.3%) of being given one of three assignments: a multi-mineral natural product (Aquamin®); a calcium-only supplement; or a placebo ("sugar pill"). Each participant will be required to take four capsules per day (two taken in the morning and two in the evening) for 90 days. Neither they nor the study team investigators will know which product they are receiving. That information will be kept in the hands of the pharmacist who dispenses the agent that participant will take.

* Each participant will be given a physical examination, which will include measurements of his/her height, weight, and vital signs (temperature, blood pressure, heart rate, breathing rate).
* The study nurse or physician's assistant will review participant's past medical history.
* Participants will be asked about any other medical conditions that they may have and all medication(s) they are currently taking. It is important that participants tell the study personnel about any medications they are taking including over-the-counter medications, calcium supplements with or without vitamin D, other vitamins, herbal medications and alternative medicines. Participants may need to stop some of their medicines in order to participate in this study. Participants are instructed to inform study personnel at any time during the study participation if they begin to take any medication(s).
* Study participants will be asked about their intake of foods and supplements containing calcium and vitamin D.
* Participants will be asked to provide information regarding their usual food that they eat (over a year), past year diet history questionnaire (DHQ II)
* Participants will be asked to take a pregnancy test within 14 days before the start of the study if she is a woman able to become pregnant.
* Participants will be asked to not take calcium, vitamin D, fiber, ginger, or fish oil supplements (including multivitamins that have low amounts) for 14 days before the study begins and for 90 days after the study begins.

Study Treatment Period (Baseline Visit through day 90) The second visit will take place within 60 days of the screening visit at the MCRU. This visit will take about 1.5 hours.

During this Baseline Visit, the following will be performed:

• Each participant will have a flexible sigmoidoscopy with colon biopsies (where twelve tissue pieces will be removed). At this time a stool sample will also be collected using the sigmoidoscope. The flexible sigmoidoscopy will be done without bowel preparations such as those used before a colonoscopy. A gastroenterologist who routinely does this procedure will do the sigmoidoscopy and remove the tissue / stool samples.

Flexible sigmoidoscopy is a test that allows the investigators to look at the inside of the colon (large intestine) from the rectum up to 15 centimeters (about 7 inches) into the colon. For the flexible sigmoidoscopy, subject will lie on its left side on the examining table. The investigator will insert a short, flexible, lighted tube into the rectum and slowly guide it into the colon. The tube is called a sigmoidoscope (sig-MOY-duh-skope). The scope transmits an image of the inside of the rectum and colon so the investigators can carefully examine the lining of participant's colon. The scope also blows air into the colon, which inflates it and helps the investigators to see better. During the flexible sigmoidoscopy, the investigator will remove several small pieces of the lining of the colon (these are called colon biopsies) using forceps instrument inserted into the scope. Each of the two sigmoidoscopy procedures (one at the beginning of the study and the other after the participant have completed taking the agent) requires twelve biopsies (5 mg each; about the size of a grain of wheat).

* Each participant will have 10 ml (or 2 teaspoons) of blood drawn from a vein.
* Each participant will be requested to give a fresh urine sample which will be collected at the beginning of this visit, before sigmoidoscopy.
* At the end of this visit (Baseline Visit), all participants will receive the assigned study agent and instructions for taking the study agent.

Between the beginning of the study treatment period and the end of the study (days 1 through 90):

Participants will take capsules containing the assigned study agent (the multi-mineral natural product or calcium or placebo) for 90 days. This will entail taking a total of four capsules per day.

The capsules should be taken as follows:

Two in the morning and two in the evening. It is suggested that they be taken at meals, but this is not required. Subjects can ingest the capsules with as much liquid that they choose.

Participants must avoid starting any new medications or supplements, such as over the counter calcium supplements (with or without vitamin D), as well as systemic (by mouth) corticosteroids such as Prednisone and Cortisol. Also, participants should not begin a course of antibiotic with any cephalosporin antibiotic including rocephin, keflex or omnicef. If participants are prescribed a cephalosporin antibiotic during the course of study, discuss this with their physician and the study team. Also, once a month each participant will receive a phone call or email from the researchers to determine whether they are experiencing any problems related to the study or any side-effects and to ask how many capsules each participant has taken. If a participant is a woman who is able to get pregnant, she must use a reliable method of birth control throughout the study. If a participant thinks she might be pregnant, she should contact the study team immediately. The study team will arrange for a pregnancy test.

End of Study Treatment Period (Final Visit) (Day 90)

Within a week after Day-90, each participant will have his/her last visit at the MCRU. This Final Visit will take about 1 hour. During the End of Study Treatment Final Visit, the following will happen:

* Participants will have a second flexible sigmoidoscopy (where twelve colon biopsies will be taken as well as stool samples).
* Participants will answer a questionnaire about whether they believed they received the Aquamin®, calcium or the placebo capsules, any untoward effects of the agents and the overall study experience.
* Participants will return any unused capsules and answer questions about any study drug they did not take.
* Each participant will have 10 ml (or 2 teaspoons) of blood drawn from a vein.
* Each participant will be requested to give a fresh urine sample which will be collected at the beginning of this visit, before sigmoidoscopy.
* Participants will tell the researchers if they had any negative reactions, side-effects, or problems over the last month of the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to give written informed consent.
* Be generally healthy, male or female, ages 18 to 80 years old.
* Must have one of the following:

  i)A first degree relative (father/mother, son/daughter, brother/sister) with colorectal cancer under the age of 60 at the time of diagnosis; OR ii)Participant have had a colorectal polyp. OR iii)Participant have previously had removed early stage colon cancer (stage I or II removed surgically and without recommendation for adjuvant therapy or with stage III colorectal cancer (CRC) treated with curative surgery >5 years ago). iv)Pre-menopausal women with intact female reproductive organs must have a negative pregnancy test within 2 weeks of the baseline flexible sigmoidoscopy. Post-menopausal is defined as no menses for the previous 12 months. If cessation of menses is within 12 months then the subject should be treated as pre-menopausal and a pregnancy test performed.

Exclusion Criteria:

* Must not be pregnant or lactating women and women of child bearing potential unwilling to use acceptable birth control throughout the study.
* Participants must not have a history or diagnosis of any of the following conditions:

  i)Kidney disease, including kidney "stones" or hypercalcemia. ii)Crohn's disease, or inflammatory bowel disease. iii)Any stomach or intestinal bleeding disorders (gastrointestinal bleeding from gastric or duodenal ulcers, or gastrin secreting tumors) or active gastric / duodenal ulcers - peptic ulcer disease (without bleeding in last 3 months). iv)Coagulopathy/hereditary hemorrhagic disorders/ or receiving therapeutic doses of Coumadin or heparin. v)Hereditary and familial polyposis (HNPCC/ familial adenomatous polyposis (FAP); Lynch Syndrome) because these are rare conditions with unique etiology.
* Participants will be excluded if they have taken the following, within the last 14 days or are unwilling to forgo the following for 14 days prior to entry into the study:

  i)Calcium, Vitamin D, ginger, or fish oil supplements, including multivitamins that have low amounts of calcium/Vitamin D and fiber supplements. ii)Non-steroidal anti-inflammatory medications (NSAIDS), such as Aspirin or Ibuprofen (except for occasional pain control or low dose aspirin for cardiovascular disease prevention). iii)Corticosteroids (a type of steroid drug such as prednisone or cortisol that helps your body to regulate your stress response, immune response and inflammation). iv)Cephalosporin antibiotics (e.g., rocephin, keflex, omnicef).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Biomarkers of Risk for Colorectal Cancer | 90 days
  A panel of biomarkers of risk for colorectal cancer in colonic mucosal biopsies of normal appearing tissue: proliferation marker (Ki67), differentiation markers (E-cadherin, AE1/AE3 and cytokeratin [CK 20]), β-catenin, extracellular calcium-sensing receptor (CaSR), Caspase-3, bax and survivin assessed by quantitative immunohistology. The purpose is to compare growth, differentiation and apoptosis biomarkers, pre and post intervention.
Colonic-mucosal Associated Microbial Profile. | 90 days
  In colonic mucosa and stool samples: Microbial analysis will be performed on colonic mucosa and stool samples. This analysis will show the difference in microbial communities before and after the intervention.
Colonic-mucosal Associated Metabolomic Profile. | 90 days
  In serum, colonic mucosa and stool samples: Metabolomic (targeted and untargeted) profile will be assessed in serum, stool and colonic mucosal biopsies. These analyses will show the difference in the metabolomic profile before and after the intervention.

SECONDARY OUTCOMES:
Biomarkers of bone turnover / metabolism. | 90 days
  In serum and urine: Serum biomarkers of bone turn-over (osteocalcin, procollagen type 1 N propeptide; P1NP , serum collagen type 1 cross-linked C-telopeptide; CTX, bone-specific alkaline phosphatase and tartrate-resistant acid phosphatase;TRAP-5b) will be assessed. Urinary collagen type 1 cross-linked N-telopeptide; NTX and urinary collagen type 1 cross-linked C-telopeptide; CTX will also be assessed pre and post intervention.
Biomarkers of liver function | 90 days
  In serum: Serum levels of hepatic enzymes; Alanine transaminase (ALT), Aspartate aminotransferase (AST) and Alkaline phosphatase (ALKP) will be assessed pre and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: James Varani, PhD, Principal Investigator — University of Michigan; Muhammad N Aslam, MD, Study Director — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Aslam MN, Bhagavathula N, Paruchuri T, Hu X, Chakrabarty S, Varani J. Growth-inhibitory effects of a mineralized extract from the red marine algae, Lithothamnion calcareum, on Ca(2+)-sensitive and Ca(2+)-resistant human colon carcinoma cells. Cancer Lett. 2009 Oct 8;283(2):186-92. doi: 10.1016/j.canlet.2009.03.037. Epub 2009 Apr 24. PMID 19394137
- [Background] Aslam MN, Paruchuri T, Bhagavathula N, Varani J. A mineral-rich red algae extract inhibits polyp formation and inflammation in the gastrointestinal tract of mice on a high-fat diet. Integr Cancer Ther. 2010 Mar;9(1):93-9. doi: 10.1177/1534735409360360. Epub 2010 Feb 11. PMID 20150219
- [Background] Aslam MN, Kreider JM, Paruchuri T, Bhagavathula N, DaSilva M, Zernicke RF, Goldstein SA, Varani J. A mineral-rich extract from the red marine algae Lithothamnion calcareum preserves bone structure and function in female mice on a Western-style diet. Calcif Tissue Int. 2010 Apr;86(4):313-24. doi: 10.1007/s00223-010-9340-9. Epub 2010 Feb 24. PMID 20180099
- [Background] Aslam MN, Bergin I, Naik M, Hampton A, Allen R, Kunkel SL, Rush H, Varani J. A multi-mineral natural product inhibits liver tumor formation in C57BL/6 mice. Biol Trace Elem Res. 2012 Jun;147(1-3):267-74. doi: 10.1007/s12011-011-9316-2. Epub 2012 Jan 6. PMID 22222483
- [Background] Attili D, Jenkins B, Aslam MN, Dame MK, Varani J. Growth control in colon epithelial cells: gadolinium enhances calcium-mediated growth regulation. Biol Trace Elem Res. 2012 Dec;150(1-3):467-76. doi: 10.1007/s12011-012-9503-9. Epub 2012 Sep 19. PMID 23008064
- [Background] Aslam MN, Bergin I, Naik M, Paruchuri T, Hampton A, Rehman M, Dame MK, Rush H, Varani J. A multimineral natural product from red marine algae reduces colon polyp formation in C57BL/6 mice. Nutr Cancer. 2012;64(7):1020-8. doi: 10.1080/01635581.2012.713160. Epub 2012 Oct 4. PMID 23035966
- [Background] Aslam MN, Bergin I, Jepsen K, Kreider JM, Graf KH, Naik M, Goldstein SA, Varani J. Preservation of bone structure and function by Lithothamnion sp. derived minerals. Biol Trace Elem Res. 2013 Dec;156(1-3):210-20. doi: 10.1007/s12011-013-9820-7. Epub 2013 Oct 6. PMID 24096551
- [Background] Dame MK, Jiang Y, Appelman HD, Copley KD, McClintock SD, Aslam MN, Attili D, Elmunzer BJ, Brenner DE, Varani J, Turgeon DK. Human colonic crypts in culture: segregation of immunochemical markers in normal versus adenoma-derived. Lab Invest. 2014 Feb;94(2):222-34. doi: 10.1038/labinvest.2013.145. Epub 2013 Dec 23. PMID 24365748
- [Background] Singh N, Aslam MN, Varani J, Chakrabarty S. Induction of calcium sensing receptor in human colon cancer cells by calcium, vitamin D and aquamin: Promotion of a more differentiated, less malignant and indolent phenotype. Mol Carcinog. 2015 Jul;54(7):543-53. doi: 10.1002/mc.22123. Epub 2013 Dec 17. PMID 26076051
- [Background] Varani J. Calcium, calcium-sensing receptor and growth control in the colonic mucosa. Histol Histopathol. 2011 Jun;26(6):769-79. doi: 10.14670/HH-26.769. PMID 21472691
- [Background] Chakrabarty S, Radjendirane V, Appelman H, Varani J. Extracellular calcium and calcium sensing receptor function in human colon carcinomas: promotion of E-cadherin expression and suppression of beta-catenin/TCF activation. Cancer Res. 2003 Jan 1;63(1):67-71. PMID 12517779
- [Background] Chakrabarty S, Wang H, Canaff L, Hendy GN, Appelman H, Varani J. Calcium sensing receptor in human colon carcinoma: interaction with Ca(2+) and 1,25-dihydroxyvitamin D(3). Cancer Res. 2005 Jan 15;65(2):493-8. PMID 15695391
- [Background] Bhagavathula N, Hanosh AW, Nerusu KC, Appelman H, Chakrabarty S, Varani J. Regulation of E-cadherin and beta-catenin by Ca2+ in colon carcinoma is dependent on calcium-sensing receptor expression and function. Int J Cancer. 2007 Oct 1;121(7):1455-62. doi: 10.1002/ijc.22858. PMID 17557293
- [Background] Aslam MN, Jepsen KJ, Khoury B, Graf KH, Varani J. Bone structure and function in male C57BL/6 mice: Effects of a high-fat Western-style diet with or without trace minerals. Bone Rep. 2016 Dec;5:141-149. doi: 10.1016/j.bonr.2016.05.002. PMID 27350956
- [Background] Aslam MN, Bassis CM, Zhang L, Zaidi S, Varani J, Bergin IL. Correction: Calcium Reduces Liver Injury in Mice on a High-Fat Diet: Alterations in Microbial and Bile Acid Profiles. PLoS One. 2017 Jan 9;12(1):e0170136. doi: 10.1371/journal.pone.0170136. eCollection 2017. PMID 28068422
- [Background] Aslam MN, Varani J: The Western-Style Diet, Calcium Deficiency and Chronic Disease Journal of Nutrition & Food Science 6(3): 496, 2016.
- [Background] McClintock SD, Colacino JA, Attili D, Dame MK, Richter A, Reddy AR, Basrur V, Rizvi AH, Turgeon DK, Varani J, Aslam MN. Calcium-Induced Differentiation of Human Colon Adenomas in Colonoid Culture: Calcium Alone versus Calcium with Additional Trace Elements. Cancer Prev Res (Phila). 2018 Jul;11(7):413-428. doi: 10.1158/1940-6207.CAPR-17-0308. Epub 2018 Apr 10. PMID 29636350
- [Background] Attili D, McClintock SD, Rizvi AH, Pandya S, Rehman H, Nadeem DM, Richter A, Thomas D, Dame MK, Turgeon DK, Varani J, Aslam MN. Calcium-induced differentiation in normal human colonoid cultures: Cell-cell / cell-matrix adhesion, barrier formation and tissue integrity. PLoS One. 2019 Apr 17;14(4):e0215122. doi: 10.1371/journal.pone.0215122. eCollection 2019. PMID 30995271
- [Background] McClintock SD, Attili D, Dame MK, Richter A, Silvestri SS, Berner MM, Bohm MS, Karpoff K, McCarthy CL, Spence JR, Varani J, Aslam MN. Differentiation of human colon tissue in culture: Effects of calcium on trans-epithelial electrical resistance and tissue cohesive properties. PLoS One. 2020 Mar 5;15(3):e0222058. doi: 10.1371/journal.pone.0222058. eCollection 2020. PMID 32134920
- [Result] Aslam MN, Bassis CM, Bergin IL, Knuver K, Zick SM, Sen A, Turgeon DK, Varani J. A Calcium-Rich Multimineral Intervention to Modulate Colonic Microbial Communities and Metabolomic Profiles in Humans: Results from a 90-Day Trial. Cancer Prev Res (Phila). 2020 Jan;13(1):101-116. doi: 10.1158/1940-6207.CAPR-19-0325. Epub 2019 Nov 26. PMID 31771942
- [Result] Aslam MN, McClintock SD, Jawad-Makki MAH, Knuver K, Ahmad HM, Basrur V, Bergin IL, Zick SM, Sen A, Turgeon DK, Varani J. A Multi-Mineral Intervention to Modulate Colonic Mucosal Protein Profile: Results from a 90-Day Trial in Human Subjects. Nutrients. 2021 Mar 14;13(3):939. doi: 10.3390/nu13030939. PMID 33799486